CLINICAL TRIAL: NCT01851408
Title: Phase 2 Study of the Combination of BAY 43-9006 (Sorafenib) and CCI-779 (Temsirolimus) in Patients With Metastatic Melanoma
Brief Title: Sorafenib and Temsirolimus in Treating Patients With Metastatic, Recurrent, or Unresectable Melanoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No progression of Phase 1 trial to Phase 2.
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000480157; 2005-0215; N01CM62202 (NIH); NCI-2009-00131 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2013-05-09; First posted 2013-05-10 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2013-05

CONDITIONS: Melanoma; Recurrent Melanoma; Stage III Melanoma; Stage IV Melanoma
Keywords: Sorafenib; Temsirolimus; Stage IV; recurrent; unresectable; non-choroidal origin; CCI-779; BAY43-9006; metastatic melanoma
MeSH Terms: conditions — Melanoma; Recurrence | interventions — Sorafenib; temsirolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temsirolimus + Sorafenib (Experimental): Temsirolimus intravenous (IV) over 30 minutes on days 1, 8,15, and 22 and oral sorafenib once or twice daily on days 1-28.
  Interventions: Drug: sorafenib tosylate; Drug: temsirolimus

INTERVENTIONS:
Drug: sorafenib tosylate — Given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Drug: temsirolimus — Given IV
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel

SUMMARY:
This phase II portion of the trial is studying the side effects and best dose of temsirolimus when given together with sorafenib and to see how well they work in treating patients with metastatic, recurrent, or unresectable melanoma. Sorafenib and temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Sorafenib may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving sorafenib together with temsirolimus may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

* To evaluate the clinical activity, in terms of overall response rate (complete and partial response), of this regimen in these patients. (Phase II)
* To evaluate the in vivo biological activity of this regimen in these patients.

SECONDARY OBJECTIVES:

I. To determine the progression-free survival and overall survival of patients treated with this regimen.

II. To determine the safety and toxicity of this regimen in these patients.

III. To Determine the population pharmacokinetics of this regimen in these patients.

IV. To correlate tumor and blood biomarkers with clinical outcome in patients treated with this regimen.

OUTLINE: Upon completion of the multicenter, phase I, dose-escalation study followed to be followed by this phase II, open-label study.

Patients receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22 and oral sorafenib once or twice daily on days 1-28. Treatment course repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3-6 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed melanoma, meeting 1 of the following criteria: recurrent or unresectable stage III disease, stage IV disease, non-choroidal origin.
* Tumor must be accessible to biopsy unless appropriate tumor sample collection has occurred within the past 3 months and patient agrees to provide these samples for this study.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Bilirubin normal
* Creatinine normal or creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 30 days after completion of study treatment.
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to sorafenib or temsirolimus.
* No uncontrolled hypertension, defined as systolic blood pressure > 140 mm Hg on 2 separate days < 1 week prior to study entry OR diastolic pressure > 90 mm Hg on 2 separate days < 1 week prior to study entry.
* No evidence of bleeding diathesis or coagulopathy.
* No condition that would impair the ability to swallow pills (e.g., gastrointestinal tract disease resulting in an inability to take oral medication; requirement for IV alimentation; or active peptic ulcer disease).
* No uncontrolled illness including, but not limited to, any of the following: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric illness or social situations that would limit study compliance.
* No traumatic injury within the past 3 weeks.
* No more than 1 prior systemic chemotherapy regimen for metastatic melanoma (Phase II).
* No prior sorafenib, temsirolimus, or any other agents targeting raf, vascular endothelial growth factor (VEGF)/VEGF receptor, or mTOR (Phase II).
* No prior surgical procedures affecting absorption.
* At least 3 weeks since prior major surgery.
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C) for melanoma and recovered.
* At least 4 weeks since prior radiotherapy and recovered.
* Prior biologic or immunotherapeutic regimens allowed.
* Prior regional chemotherapy regimens (e.g., isolated limb perfusion) allowed but only 1 prior regional chemotherapy regimen allowed if all target lesions are within the prior regional treatment field.
* No concurrent enzyme-inducing antiepileptic drugs including, but not limited to, any of the following: phenytoin, carbamazepine, phenobarbital, rifampin or Hypericum perforatum (St. John's wort).
* No concurrent prophylactic hematopoietic colony-stimulating factors.
* No other concurrent investigational agents.
* No other concurrent anticancer agents or therapies for this cancer.
* No concurrent full-dose anticoagulation (i.e., warfarin, IV heparin, or low-molecular weight heparin).
* No concurrent grapefruit or grapefruit juice.
* No concurrent combination antiretroviral therapy for HIV-positive patients.
* Concurrent prophylactic anticoagulation therapy (e.g., low-dose warfarin) allowed provided prothrombin time (PT) international normalized ratio (INR) < 1.1 times upper limits of normal (ULN).
* Unidimensionally measurable disease >= 20 mm by conventional techniques or >= 10 mm by spiral computed tomography (CT) scan (longest diameter to be recorded) and margins of visible cutaneous metastatic lesions should be clearly defined and measured in at least one dimension as >= 10 mm.
* No known brain metastases unless the following criteria are met: no radiographical evidence of recurrences in the brain >= 3 months after complete resection of the brain metastases, asymptomatic brain metastases stable for >= 3 months since whole-brain radiation therapy and/or stereotactic radiosurgery and must not require steroid for brain metastases.
* White Blood Count (WBC) >= 3,000/mm³
* Absolute neutrophil count >= 1,500/mm³
* Platelet count >= 100,000/mm³
* Serum cholesterol =< 350 mg/dL
* Triglycerides =< 400 mg/dL
* Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) =< 2.5 times upper limit of normal.
* No peripheral neuropathy > grade 2.
* At least 5 years since prior chemotherapy for other types of cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Objective response rate (complete response and partial response) CCI-779 in combination with BAY43-9006 | Up to 5 years

SECONDARY OUTCOMES:
Progression-free survival | The duration of time from start of treatment to date of first evidence of progression or the date of last follow-up for patients who do not progress, assessed up to 5 years
  Kaplan-Meier life table methods and Cox proportional hazards regression modeling will be utilized to analyze progression-free survival and overall survival.
Overall survival | 5 years
  Kaplan-Meier life table methods and Cox proportional hazards regression modeling will be utilized to analyze progression-free survival and overall survival.
Noncompartmental pharmacokinetic parameters of BAY43-9006 and CCI-779 estimated using a validated commercial software | Week 1 and 3
  Maximum concentration (Cmax) and time to Cmax (tmax) will be the observed values. Area under the plasma concentration-time curve from zero to last observable time (AUClast).

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Kim, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center official website — http://www.mdanderson.org